CLINICAL TRIAL: NCT04628143
Title: Open-label, Multi-center, Randomized Controlled, Phase 2 Clinical Trial to Evaluate the Efficacy and Safety of CKD-314 in Hospitalized Adult Patients Diagnosed With COVID-19
Brief Title: A Study Evaluating the Efficacy and Safety of CKD-314 in Hospitalized Adult Patients Diagnosed With COVID-19 Pneumonia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A108_01CVD2013
Record Dates: First submitted 2020-11-10; First posted 2020-11-13 (Actual); Last update posted 2021-08-13 (Actual); Status verified 2021-04

CONDITIONS: COVID-19
Keywords: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — nafamostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (No Intervention): Standard of Care Treatment for COVID-19 Infection
- Nafamostat + Standard of Care (Experimental): Nafamostat mesylate on top of standard of care
  Interventions: Drug: Nafamostat Mesilate

INTERVENTIONS:
Drug: Nafamostat Mesilate — Administered intravenously as a continuous infusion
  Other Names: CKD-314
  Arms: Nafamostat + Standard of Care

SUMMARY:
The primary objective of this study is to evaluate the efficacy of CKD-314 (Nafabelltan) compared to standard of care (SOC), with respect to clinical status assessed by a 7-point ordinal scale in hospitalized adult patients diagnosed with COVID-19 pneumonia

DETAILED DESCRIPTION:
Open-label, Multi-center, Randomized Controlled, Phase 2 Clinical Trial to Evaluate the Efficacy and Safety of CKD-314 in Hospitalized Adult Patients Diagnosed with COVID-19

ELIGIBILITY:
Inclusion Criteria:

* Men and women Aged ≥18 years
* Hospitalized subjects who have confirmed COVID-19 infection and have evidence of pneumonia:

  * COVID-19 infection: SARS-CoV-2 positive confirmed by RT-PCR

    * Pneumonia: A reliable diagnosis of new lung infiltration on a chest CT scan or chest radiograph
* Subjects within 72 hours after confirmed COVID-19 pneumonia
* Subjects with a seven-category ordinal scale of clinical status of 4 (hospitalization, requiring supplemental oxygen) or 5 (hospitalization, requiring nasal high-flow oxygen therapy and/or noninvasive mechanical ventilation)
* Subjects (or legally authorized representative) should be able to understand and agree to comply with the clinical trial and to provide a written consent document prior to initiation of any study procedure

Exclusion Criteria:

* Subject has a serious chronic disease
* Subject requiring invasive mechanical ventilation at the time of screening
* Subject with rapidly(within 3 days) deteriorating clinical condition according to the investigator's opinion
* Subject who have a record of HIV or AIDS
* Subject taking corticosteroids[However, ① steroids being used for the treatment of Corona 19 (eg, Dexamethasone, etc.), ② topical steroids,

  ③ Patients who are administering inhaled steroids are not eligible for exclusion]
* Subject taking immunosuppressants/immunomodulators
* Subject with liver cirrhosis whose Child-Pugh score is B or C
* Subject with hyperkalemia (K> 5.1mmol/L)
* Subject who have liver disease abnormalities with ALT or AST > 5 times ULN
* Estimated glomerular filtration rate (eGFR) < 30 ml/min
* QTc >500ms
* Subject who have hypersensitivity to the investigational drug
* Pregnant or lactating females
* Subject who are not appropriate for the study, as the investigator's opinion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2020-12-21 (Actual); Primary Completion 2021-04-05 (Actual); Study Completion 2021-04-05 (Actual)

PRIMARY OUTCOMES:
Time to clinical improvement | up to 28 days
  Time to clinical improvement (TTCI) was defined as time (days) from randomization to a decline of 2 categories on the seven-category ordinal scale of clinical status or live discharge from the hospital, whichever came first

SECONDARY OUTCOMES:
Time to recovery | up to 28 days
  Day of recovery is defined as the first day on which the subject satisfies one of the following: 1) Not hospitalized with resumption of normal activities; 2) Not hospitalized, but unable to resume normal activities; 3) Hospitalization, not requiring supplemental oxygen- no longer required ongoing medical care
Proportion of patients with clinical improvement as defined by live discharge from hospital or a decline of 2 categories on the seven-category ordinal scale of clinical status | Day 4, 7, 10, 14, 21 and 28
  Proportion of patients with clinical improvement as defined by live discharge from hospital or a decline of 2 categories on the seven-category ordinal scale of clinical status

CONTACTS AND LOCATIONS:
Overall Officials: Dongho Kim, MD, Principal Investigator — Korea Cancer Center Hospital
Locations (1):
- Korea Cancer Center Hospital, Seoul, South Korea